CLINICAL TRIAL: NCT04501354
Title: Evaluation of Clinical and Bone Density Improvement After Implantation of Allogenic Mesenchymal Stem Cell From Umbilical Cord on Osteoporosis Patients (Clinical Trial)
Brief Title: Evaluation of Clinical and Bone Density Improvement After Implantation of Allogenic Mesenchymal Stem Cell From Umbilical Cord on Osteoporosis Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahmad Jabir Rahyussalim (Other)
Responsible Party: Sponsor-Investigator, Ahmad Jabir Rahyussalim, Orthopaedic and Traumatology Specialist, Principal Investigator, Indonesia University
Organization: Indonesia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-08-1018
Record Dates: First submitted 2020-08-02; First posted 2020-08-06 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UC-Mesenchymal Stem Cell (Experimental): Allogeneic Mesenchymal Stem Cell from umbilical cord
  Interventions: Drug: Mesenchymal Stem Cell

INTERVENTIONS:
Drug: Mesenchymal Stem Cell — Mesenchymal Stem Cell + NaCl 0,9% 2ml

SUMMARY:
This study will assess the effectiveness of the allogeneic mesenchymal cell from umbilical cord in improving the quality and quantity of spinal density of osteoporosis patients proven by the results of Bone Mass Density (BMD) examination compared to baseline and evaluate improvement of quality of pain with visual analog scale (VAS).

DETAILED DESCRIPTION:
Currently, preventive and therapeutic strategies for osteoporosis patients are based on calcium and vitamin D supplementation, the use of pharmacological agents that inhibit bone resorption such as bisphosphonates, and sometimes calcitonin. Although bisphosphonates have been found to reduce osteoporosis, clinical use for these drugs has been limited because of its potential to produce serious side effects, such as mandibular osteonecrosis and atypical femoral fractures. Therefore, new therapeutic strategies for osteoporosis are needed.

This study will assess the effectiveness of the allogeneic mesenchymal cell from umbilical cord. Patients who have received mesenchymal stem cell therapy (MSC) are expected to have positive effects such as reduced pain sensation in the back assessed by Visual Analog Scale (VAS), improvement in the range of motion (ROM), improving the quality of osteoporosis patients's bone proven by the results of Bone Mass Density (BMD) and improvement in patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients older than 50 yrs old.
2. Female patients older than 40 years old.
3. Patients enrolled in Cipto Mangunkusumo Hospital with osteoporosis confirmed by BMD test.
4. Patients with no history of autoimun disease (SLE, Addison's disease, Chron's disease) and other diseases related to osteoporosis.
5. Patients with no history of consuming drug related osteoporosis.
6. No active infection confirmed by HbsAg, HIV, CMV, Rubella and Toxoplasma examination.
7. Agree to participate the study by signing informed consent form.

Exclusion Criteria:

1. Patients with autoimun diesasde (SLE, Addison's diesase, Chron's disease and other osteoporosis related disease.
2. Patients under immunosuppressive, anticoagulant or corticosteroid treatment.
3. Paralysis patients after surgical treatment
4. Patients under 20 years old
5. Declined to participate in the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 5 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Bone Mass Density (BMD) | 6 months
  Improvement of spinal density in osteoporosis patients proven by the results of Bone Mass Density (BMD).
  1. Above Standard Deviation (SD) (-1) means normal
  2. Between SD (-1) and (-2.5) is classified as osteopenia. Osteopenia is a condition when bone density is lower than the average, but not as low as osteoporosis.
  3. Below SD (-2.5) is categorized as osteoporosis.
  The numbers are expected to be higher after MSC implantation.
Visual Analog Scale (VAS) | 6 months
  Evaluates pain quality using Visual Analog Scale (VAS) from 0 - 10. Zero is no pain at all, one is the the least pain and ten is the most painful. The numbers are expected to be lower after MSC implantation.

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia